CLINICAL TRIAL: NCT02645409
Title: Intraoperative Folate Targeted Fluorescence in Renal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chandru Sundaram (Other)
Responsible Party: Sponsor-Investigator, Chandru Sundaram, Professor, Director of the Residency Program and Minimally Invasive Surgery, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0546
Record Dates: First submitted 2015-12-08; First posted 2016-01-01 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Fluorescence; Imaging; Partial nephrectomy; Radical nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Partial nephrectomy (Experimental): OTL38 will be given approximately 2 hours before surgery. Intraoperative fluorescent imaging will utilized in parallel with standard operating procedures for partial nephrectomy. Photographs of the surgery field and tumor (ex-vivo) will be taken under normal light and fluorescent light.
  Interventions: Drug: OTL38; Device: Intraoperative fluorescence imaging system
- Radical nephrectomy (Experimental): OTL38 will be given approximately 2 hours before surgery. Intraoperative fluorescent imaging will utilized in parallel with standard operating procedures for radical nephrectomy. Photographs of the surgery field and tumor (ex-vivo) will be taken under normal light and fluorescent light.
  Interventions: Drug: OTL38; Device: Intraoperative fluorescence imaging system

INTERVENTIONS:
Drug: OTL38 — OTL38 is a folate analog conjugated with a fluorescent dye that emits light in the near infrared spectrum. This longer wavelength allows for deeper penetration of the fluorescent light through tissues with the potential to better image tumors beneath adipose tissue or deeper into organ parenchyma.
Device: Intraoperative fluorescence imaging system

SUMMARY:
Primary

• To explore the use of OTL38 and fluorescence imaging to detect RCC in partial nephrectomy at the margins of resection, and in lymph node(s) or other metastases during radical nephrectomy.

DETAILED DESCRIPTION:
Administration of the study drug, OTL38, will begin prior to skin incision in the preoperative area where safety monitoring will occur. The tumor resection occurs approximately 2 hours after being brought back to the operating room and so there is no wait time between infusion and being taken back to operating room. Intraoperative fluorescent imaging will be utilized in parallel with the standard operating procedure to capture images during surgery. Images also will be taken of the excised specimen on the back table. The excised specimen will be sent to the pathology department for fluorescent imaging and immunohistochemistry for FR. Subjects will have a 2-5 day hospital stay (normal nephrectomy recovery period) where safety measurements will be taken. Final safety measurements will be taken at the 10-day and 1-month follow-up visits.

ELIGIBILITY:
Inclusion criteria for localized RCC treated with partial nephrectomy

To be considered eligible to participate in this study, a patient must meet all the inclusion criteria listed below:

* ≥ 18 years of age.
* Have primary or suspected diagnosis of RCC, with presence of cT1-2 renal mass by diagnostic CT assessment.
* Scheduled for partial nephrectomy of renal mass.
* Expected survival of at least 3 months.
* Written informed consent available.
* ECOG ≤ 1 (Appendix G).
* Negative serum or urine pregnancy test within 24 hours for females of child bearing age
* Recovered from toxicity of any prior therapy to ≥ grade 1.

Inclusion criteria for advanced RCC treated with radical nephrectomy

To be considered eligible to participate in this study, a patient must meet all the inclusion criteria listed below:

* ≥ 18 years of age.
* Have pathologic or suspected diagnosis of RCC with presence of cT1-4 renal mass and evidence of nodal or metastatic involvement by diagnostic CT assessment
* Scheduled for radical nephrectomy and lymph node dissection.
* Expected survival of at least 3 months.
* ECOG ≤ 2.
* Negative serum or urine pregnancy test within 24 hours for females of child bearing age.
* Recovered from toxicity of any prior therapy to ≥ grade 1
* Written informed consent available.

Exclusion criteria for both localized and advanced RCC

* History of any anaphylactic reaction, any severe allergy, or any allergy to folate.
* Brain metastases
* Baseline GFR < 50 mL/min/1.73m2)
* Hepatic toxicity ≥ Grade 2 (using CTCAE version 4 standard definitions).
* Participation in another investigational drug trial either concurrently or 30 days prior to surgery
* Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient, limit the patient's ability to complete the study, and/or compromise the objectives of the study.
* Known sensitivity to fluorescent light

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandru P. Sundaram, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Partial Nephrectomy: OTL38 will be given approximately 2 hours before surgery. Intraoperative fluorescent imaging will utilized in parallel with standard operating procedures for partial nephrectomy. Photographs of the surgery field and tumor (ex-vivo) will be taken under normal light and fluorescent light.
  OTL38: OTL38 is a folate analog conjugated with a fluorescent dye that emits light in the near infrared spectrum. This longer wavelength allows for deeper penetration of the fluorescent light through tissues with the potential to better image tumors beneath adipose tissue or deeper into organ parenchyma.
  Intraoperative fluorescence imaging system
Period: Overall Study
Arm/Group | Partial Nephrectomy | Radical Nephrectomy
Started | 14 | 0 (It was decided to not continue with the Radical Nephrectomy arm of the study.)
Completed | 10 | 0
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The protocol was amended to stop at the partial nephrectomy arm because the equipment needed for the radical nephrectomy arm was only for open surgery as opposed to robotic or laparoscopic surgery which is the preferred method for the PI.
Groups:
- Radical Nephrectomy: OTL38 will be given approximately 2 hours before surgery. Intraoperative fluorescent imaging will utilized in parallel with standard operating procedures for radical nephrectomy. Photographs of the surgery field and tumor (ex-vivo) will be taken under normal light and fluorescent light.
  OTL38 is a folate analog conjugated with a fluorescent dye that emits light in the near infrared spectrum. This longer wavelength allows for deeper penetration of the fluorescent light through tissues with the potential to better image tumors beneath adipose tissue or deeper into organ parenchyma.
- Total: Total of all reporting groups
Arm/Group | Partial Nephrectomy | Radical Nephrectomy | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Customized [Count of Participants; unit: Participants]
  50-70 | 10 |  | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 9 |  | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 10 |  | 10
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 |  | 10
BMI [Mean (Full Range); unit: kg/m^2] | 29.4 [23.2 to 34.4] |  | 29.4 [23.2 to 34.4]
Pathologic Tumor Stage [Count of Participants; unit: Participants]
  pT1a | 8 |  | 8
  pT3a | 1 |  | 1
  Benign | 1 |  | 1
Negative Post-Surgical Margins [Count of Participants; unit: Participants] — Negative post-surgical margins means that no cancer cells were identified at the edge of the tissue.
  Participants | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Fluorescence of cT1 RCC in Partial Nephrectomy Specimens
Description: Pathology results will be compared with immunohistochemistry results for each patient. Fluorescence will be looked for in the margins of resection for partial nephectomy and in regional lymph nodes and metastases for radical nephrectomy.
Time Frame: During procedure, an average of 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Nephrectomy
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 30 days
Description: There are zero participants at risk in the radical nephrectomy arm because no patients enrolled in this arm
Groups:
- Radical Nephrectomy: OTL38 is a folate analog conjugated with a fluorescent dye that emits light in the near infrared spectrum. This longer wavelength allows for deeper penetration of the fluorescent light through tissues with the potential to better image tumors beneath adipose tissue or deeper into organ parenchyma.
  OTL38 is a folate analog conjugated with a fluorescent dye that emits light in the near infrared spectrum. This longer wavelength allows for deeper penetration of the fluorescent light through tissues with the potential to better image tumors beneath adipose tissue or deeper into organ parenchyma
Arm/Group | Partial Nephrectomy | Radical Nephrectomy
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 1/10 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial Nephrectomy (N=10) | Radical Nephrectomy (N=0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02645409/Prot_SAP_000.pdf